CLINICAL TRIAL: NCT00376922
Title: Use of Music to Reduce Anxiety & Perceived Pain for Adult Patients With Hematological Malignancies Undergoing Bone Marrow Biopsy
Brief Title: Music in Reducing Anxiety and Pain in Adult Patients Undergoing Bone Marrow Biopsy for Hematologic Cancers or Other Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000495315; CCCWFU-98306; CCCWFU-IRB00000468
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2012-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Pain; Precancerous Condition; Psychosocial Effects of Cancer and Its Treatment
Keywords: pain; psychosocial effects of cancer and its treatment; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; essential thrombocythemia; extramedullary plasmacytoma; meningeal chronic myelogenous leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; polycythemia vera; previously treated myelodysplastic syndromes; primary systemic amyloidosis; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage III multiple myeloma; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; mast cell leukemia; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; T-cell large granular lymphocyte leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; refractory hairy cell leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; untreated hairy cell leukemia; recurrent adult Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; adult grade III lymphomatoid granulomatosis; recurrent adult grade III lymphomatoid granulomatosis; Waldenström macroglobulinemia; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; recurrent adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; recurrent adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; contiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; isolated plasmacytoma of bone; monoclonal gammopathy of undetermined significance; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; post-transplant lymphoproliferative disorder; primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Pain; Precancerous Conditions; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Thrombocythemia, Essential; Polycythemia Vera; Immunoglobulin Light-chain Amyloidosis; Leukemia, Prolymphocytic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Mast-Cell; Leukemia, Large Granular Lymphocytic; Leukemia, Hairy Cell; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Monoclonal Gammopathy of Undetermined Significance | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care (No Intervention)
- Music therapy (Experimental)
  Interventions: Procedure: music therapy

INTERVENTIONS:
Procedure: music therapy — music played for patient during bone marrow biopsy collection
  Arms: Music therapy

SUMMARY:
RATIONALE: Listening to relaxing music during a bone marrow biopsy may be effective in reducing anxiety and pain.

PURPOSE: This randomized clinical trial is studying how well music works in reducing anxiety and pain in adult patients undergoing bone marrow biopsy for hematologic cancers or other diseases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of using music as an intervention to reduce anxiety and perceived pain in adult patients who are undergoing bone marrow biopsy for hematologic cancers or other diseases.
* Compare differences in state anxiety and perceived pain level between patients treated with or without music intervention.

OUTLINE: This is a randomized, feasibility study. Patients are stratified according to the practitioner performing the procedure. Patients are randomized to 1 of 2 treatment arms.

* Arm I (music intervention): Patients complete baseline questionnaires that measure anxiety and anticipated pain prior to bone marrow biopsy (BMB). Patients also provide demographic and clinical information, including pre-procedure medications and previous BMB experience. Patients then choose from music compact discs with various types of relaxing music (e.g., classical, country, soft rock, and R&B) and listen to the music through headphones during the bone marrow biopsy for approximately 30 minutes. After the biopsy, patients complete questionnaires that measure their response to the music, in terms of anxiety and perceived pain experienced during the procedure, and their overall level of satisfaction.
* Arm II (usual care [control]): Patients complete pre-procedure questionnaires, as in arm I, and undergo BMB without music intervention. Post-procedure questionnaires assess patient response to BMB in the absence of music and their level of satisfaction with the procedure.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hematologic malignancy
* Referred or scheduled for a bone marrow biopsy

PATIENT CHARACTERISTICS:

* Must understand written and spoken English

PRIOR CONCURRENT THERAPY:

* Prior bone marrow biopsies allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
State anxiety as measured by the State-Trait Anxiety Inventory (STAI) questionnaire | day 1
Perceived pain level as measured by the Visual Analogue Scale | day 1
Patient satisfaction as measured by a post-procedure questionnaire | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C. Danhauer, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States